CLINICAL TRIAL: NCT03076645
Title: Measure of Engagement of Epilepsy Patients in Messaging Groups and Group Characteristics That Influence Engagement.
Brief Title: Measure of Engagement of Epilepsy Patients in Messaging Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Abbas Hasan, Honorary Researcher, Royal Free Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 203594
Record Dates: First submitted 2017-02-02; First posted 2017-03-10 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): The Experimental Group will be placed in a group using the matching algorithm. Facilitator support and education intervention
  Interventions: Behavioral: Facilitator support and education

INTERVENTIONS:
Behavioral: Facilitator support and education — Group engaged with facilitator support and education

SUMMARY:
This study will measure the engagement of people with epilepsy in a mobile phone based messaging platform as well as understand if there is an impact on their self-management

DETAILED DESCRIPTION:
The primary purpose of this study is to assess a person with epilepsy's level of usage of a mobile messaging application for peer support. The secondary purpose is to understand what characteristics of their group drive different levels of usage and improvements in self-management.

Participants can participate as much or little as they want for a minimum of six weeks. Participants will complete an initial and a final questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age, diagnosis of epilepsy, have access to a smartphone capable of running messaging application

Exclusion Criteria:

* A diagnosis of learning disability/difficulty, significant mental health conditions; those in care, bereaved, or prisoners. Any other vulnerable individuals (individuals unable to protect themselves against significant harm or exploitation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Engagement | 6 weeks
  Average participant number of posts over time frame assessed by tracking number of participant entries

SECONDARY OUTCOMES:
Epilepsy self-management | Change in Baseline to 6 weeks
  Patient activation measure based on self-reported questionnaire
Epilepsy medication adherence | Change in Baseline to 6 weeks
  Medication adherence based on self-reported questionnaire
Epilepsy quality of life | Change in Baseline to 6 weeks
  Quality of life in epilepsy metric based on self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Adina Nash, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Lewisham & Greenwich NHS Trust, Lewisham
  - Barts and The London NHS Trust, London
  - Royal Free Hospital, London
  - National Hospital for Neurology and Neurosurgery, London
  - Kent Community Health NHS Trust, Maidstone

IPD SHARING:
Plan to Share IPD: No
No current resource to share individual participant data. Data will be destroyed per protocol after due course and completion of study